CLINICAL TRIAL: NCT01997086
Title: Percutaneous Transforaminal Endoscopic Discectomy (PTED) Versus Microendoscopic Discectomy (MED) for the Treatment of Lumbar Disc Herniation: A Prospective Randomized Controlled Study
Brief Title: Percutaneous Transforaminal Endoscopic Discectomy vs Microendoscopic Discectomy for Treatment of Lumbar Disc Herniation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Limin Rong, Prof., M.D., Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTED-MED
Record Dates: First submitted 2013-11-14; First posted 2013-11-27 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Lumbar Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transforaminal discectomy (Active Comparator): patients diagnosed as lumbar disc herniation undergoing percutaneous transforaminal endoscopic discectomy (PTED).
  Interventions: Procedure: Percutaneous transforaminal endoscopic discectomy (PTED)
- Microendoscopic discectomy (Active Comparator): Patients diagnosed as lumbar disc herniation undergoing microendoscopic discectomy (MED).
  Interventions: Procedure: Microendoscopic discectomy (MED)

INTERVENTIONS:
Procedure: Percutaneous transforaminal endoscopic discectomy (PTED) — Percutaneous transforaminal endoscopic discectomy
  Arms: Transforaminal discectomy
Procedure: Microendoscopic discectomy (MED) — Microendoscopic discectomy
  Arms: Microendoscopic discectomy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of two minimal invasive endoscopic discectomy, PTED and MED, for the treatment of symptomatic lumbar disc herniation.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a common pathological process leading to spinal surgery. Open discectomy used to be a widespread procedure for surgical treatment for symptomatic LDH. Currently, with rapid progress of endoscopic techniques, several minimal invasive endoscopic surgeries have been developed to perform discectomy. Percutaneous transforaminal endoscopic discectomy (PTED) and microendoscopic discectomy (MED) are two widely used minimal invasive surgical procedures, the effectiveness of which has been proved to be comparable to conventional open discectomy. As difference in operative approaches and iatrogenic injury, the clinical outcome might be dramatically different from each other.

In this study, a single center randomized controlled trial will be performed to evaluate the effectiveness of two minimal invasive endoscopic discectomy, PTED and MED, for the treatment of symptomatic LDH. We will conduct the study at the 3rd affiliated hospitals of Sun Yat-Sen University.

Two groups of patients will be investigated; 1) patients diagnosed with lumbar disc herniation undergoing PTED, and 2) patients diagnosed with lumbar disc herniation undergoing MED.

The primary outcomes of the study will be score of Oswestry Disability Index (ODI) as measured at pre- and post-operation, 1 month, 3 months, 6 months, and annually thereafter. Secondary outcomes include Visual Analog Scale (VAS), the SF-36 Health Survey, as well as post-operative radiological assessment. Treatment effect is defined as the difference in the mean change from baseline between the two groups. Lumbar intervertebral disc tissue would be obtained during surgery for histological analysis, in order to evaluate disc degeneration and find out risk factors of it.

On the basis of the results of this trial we will, for the first time, have scientific evidence as to the relative effectiveness of PTED versus MED for minimal invasive surgical treatment for symptomatic lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Persistent radicular pain.
* Signs including evidence of nerve root compression with a positive nerve root tension sign (straight leg raising test or femoral tension sign) or a corresponding sign of neurological deficit (asymmetrical depressed reflex, decreased sensation in a dermatomal distribution, or weakness in a myotomal distribution).
* An imaging study (MRI or CT) showing LDH at a level and side corresponding to the patients radicular signs or symptoms.

Exclusion Criteria:

* <18 or >65 years of age
* Insufficient conservative treatment (6 weeks)
* Cauda equina syndrome or progressive neurologic deficit requiring urgent surgical intervention
* Combination with other spinal disorder requiring advanced surgery (such as lumbar stenosis, spondylolisthesis, deformity, fracture, infection, tumor and so on)
* Equal to or more than two responsible level
* High-grade migrated disc herniation
* Previous spinal surgery
* Possible pregnancy or other comorbid conditions contraindicating surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2013-10; Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Changes in pain and functional status as measured by Oswestry Low Back Disability Questionnaire (Oswestry Disability Index,ODI) | Baseline, post-operation, 1 month, 3 months, 6 months, and annually thereafter

SECONDARY OUTCOMES:
Changes in health-related quality of life as measured by the EQ-5D,Visual Analog Scale (VAS) and the SF-36 health status questionnaire, and the radiological changes in spine as measured by x-ray, CT or MRI. | Baseline, post-op 1 month, 3 months, 6 months, and annually thereafter.
Histological analysis of surgical lumbar intervertebral disc tissue | postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Limin Rong, M.D., Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen Z, He L, Di J, Huang L, Feng F, Yang B, Xie P, Rong L. Lumbar facet joint osteoarthritis as the underlying reason for persistent low back pain after minimally invasive discectomy. Arch Orthop Trauma Surg. 2023 Jul;143(7):3811-3821. doi: 10.1007/s00402-022-04595-y. Epub 2022 Sep 17. PMID 36114871
- [Derived] Chen Z, Zhang L, Dong J, Xie P, Liu B, Chen R, Li S, Liu Z, Yang B, Feng F, He L, Yang Y, Pang M, Rong L. Percutaneous Transforaminal Endoscopic Discectomy Versus Microendoscopic Discectomy for Lumbar Disk Herniation: Five-year Results of a Randomized Controlled Trial. Spine (Phila Pa 1976). 2023 Jan 15;48(2):79-88. doi: 10.1097/BRS.0000000000004468. Epub 2022 Sep 7. PMID 36083850
- [Derived] Chen Z, He L, Huang L, Liu Z, Dong J, Liu B, Chen R, Zhang L, Xie P, Rong L. Risk Factors for Poor Outcomes Following Minimally Invasive Discectomy: A Post Hoc Subgroup Analysis of 2-Year Follow-up Prospective Data. Neurospine. 2022 Mar;19(1):224-235. doi: 10.14245/ns.2143084.542. Epub 2022 Mar 31. PMID 35378590
- [Derived] Chen Z, Zhang L, Dong J, Xie P, Liu B, Wang Q, Chen R, Feng F, Yang B, Shu T, Li S, Yang Y, He L, Pang M, Rong L. Percutaneous transforaminal endoscopic discectomy compared with microendoscopic discectomy for lumbar disc herniation: 1-year results of an ongoing randomized controlled trial. J Neurosurg Spine. 2018 Mar;28(3):300-310. doi: 10.3171/2017.7.SPINE161434. Epub 2018 Jan 5. PMID 29303469